CLINICAL TRIAL: NCT05416151
Title: Evaluation of the Effect of a 28-day B.Lactis Consumption Twice Daily on Gastro-Intestinal (GI) Symptoms in Healthy Women Reporting Minor GI Symptoms. A Proof of Efficacy, Randomized, Controlled, Double-blind, Parallel Arms, Adaptive Design.
Brief Title: Effect of B.Lactis Consumption on Gastro-Intestinal (GI) Symptoms in Healthy Women Reporting Minor GI Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NU390
Record Dates: First submitted 2022-05-12; First posted 2022-06-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Gastro-intestinal Symptoms in Healthy Subjects
Keywords: Gastro intestinal symptoms; Healthy women; Freeze-dried probiotic product; Randomized controlled trial
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: A proof-of-efficacy, randomized, controlled, double-blind, monocentric, parallel arms design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study Test and Control products have similar appearance including packaging and texture, smell, and taste, in order to preserve the double-blind methodology.
  The blinding of study products will be performed by assigning a study product number corresponding to the randomization list. Then blinded study product packages will be carried to the investigational site for assignment to the subjects.
  Product allocation will be performed by randomized method (IWRS validated system) as it is a Randomized Controlled Trial. The participants are thus assigned to intervention groups randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1, Test: freeze-dried B. lactis (Other)
  Interventions: Other: Freeze-dried biotic
- Arm 2, Control: freeze-dried maltodextrin (Other)
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Freeze-dried biotic — 2 sticks of 3g consumed daily for 28 days
  Arms: Arm 1, Test: freeze-dried B. lactis
Other: Maltodextrin — 2 sticks of 3g consumed daily for 28 days
  Arms: Arm 2, Control: freeze-dried maltodextrin

SUMMARY:
The purpose of this study is to assess the effect of a 28-day B.lactis consumption twice daily on Gastro-Intestinal (GI) symptoms in healthy women reporting minor GI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent SI01: Free-living Participant who fully understands and agree to the objectives of the study, who gave signed and dated informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Age SI02: Women between the ages of 18 and 60 years (bounds included), at the time of signing the informed consent at the inclusion visit.
* Weight SI03: Subject with body mass index (BMI) between 18.0 and 30.0 kg/m2 (bounds included).
* Type of Participant and Disease Characteristics SI04: Subject with minor digestive symptoms as defined by composite score between 12 and 16 (bounds included) or at least one digestive symptom with a score ≥4 according to the screening questionnaire of frequency of digestive symptoms (DSFQ (R)).

SI05: Subject with mean stool frequency between 3 and 21 bowel movements per week during the past month (bounds included) according to the screening questionnaire (DSFQ (R)).

* Sex SI06: Women of childbearing potential must be using a medically approved method of contraception (Oral birth control pills, Intra-uterine device (IUD) or Double barrier methods (such as condoms and spermicide)) OR women must be postmenopausal for at least 12 months prior to study entry OR women surgically sterile (i.e. hysterectomy, bilateral oophorectomy or bilateral tubal ligation).
* Other SI07: Subject willing to strictly follow dietary instructions (unauthorized products) for the entire duration of the study.

SI08: Subject must have access to adequate space to store the investigational products (storage at 4°C) and the stools samples (storage in freezer) according to the labels' storage recommendations.

SI09: Subject able to communicate well with the investigator and to comply with the requirements for the entire study.

SI10: Subject covered by health insurance or covered by a similar system. SI11: Subject agrees to be registered in the National biomedical research file for volunteers.

SI12: Subject willing to complete ePRO through a smartphone compatible with playstore or apple store and having access to internet.

Exclusion Criteria:

- Medical Conditions and History SE01: Pregnant women based on pregnancy test or planning to become pregnant during the study's participation or lactating women.

SE02: Subject with disorder of gut brain interactions according to ROME IV criteria (Functional Bowel Disorders/FBD module, Functional Dyspepsia/FD module).

SE03: Subject with gastrointestinal disorders other than minor digestive symptoms as defined in SI04 according to investigator's medical assessment.

SE04: Subject who have consulted for gastrointestinal disorders within 6 months prior to the screening visit (V1).

SE05: Subject who had any dental surgery within the last 4 weeks, or who plans to have one during the study, excluding care of tooth decay.

SE06: Subject with any antecedents of digestive surgery (except for appendectomy and cholecystectomy performed more than 2 years ago).

SE07: Subject with previous history of drug or alcohol abuse 6 months prior to screening.

SE08: Subject with severe disease as assessed by the investigator (e.g inflammatory bowel disease, benign or malign tumor of intestine or colon cancer, severe heart disease, kidney disease, neurological disease or psychiatric disease, immunodeficiency disorder).

- Prior/Concomitant Therapy SE09: Subject with any intake of antibiotics or intestinal antiseptics in the previous 2 months (within 60 days) prior to the screening visit (V1).

SE10: Subject with any intake of drugs that might modify gastrointestinal function (e.g regular use of laxatives, anti-diarrhea, prokinetics, proton pump inhibitors (PPIs)) in the previous 2 weeks (within 14 days) prior to the screening visit (V1).

SE11: Subject with any intake of over-the-counter yeasts or probiotics supplements (such as pills, tablets, sachets or sticks) in the previous 2 weeks (within 14 days) prior to the screening visit (V1).

SE12: Subject who underwent a general anesthesia in the preceding 4 weeks. SE13: Subject with known allergy to study products component (maltodextrin for example).

SE14: Subject with any current use of any medication with potential central nervous system effects as judged by the investigator (including but not limited to opiate pain medication).

- Prior/Concurrent Clinical Study Experience SE15: Subject who has planned to participate in another investigational study during the period of this study OR subject involved in any other clinical study within the preceding month except for non-investigational procedures (e.g: CT scan, endoscopy capsule) OR subject in the exclusion period after participation in another clinical study.

Diet SE16: Change of dietary habits within the 4 weeks preceding the V1 (for instance start of a diet rich in fiber) or planned change (for example to start a new diet during the study's participation).

- Other Exclusions SE17: Vulnerable subjects defined as individuals whose willingness to volunteer in the clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (examples are members of a group with a hierarchical structure linked to the Investigator or to the Sponsor, such as medical, pharmacy, dental and nursing students, subordinate hospital and laboratory personnel, employees of the Investigator or of the Sponsor, members of the armed forces, and persons kept in detention).

SE18: Subject under guardianship or curatorship. SE19: Subject expected to be living in the same home as a subject currently participating to the present study (or willing to) and to concomitantly receive some study products.

SE20: Subject planning to start or quit smoking during the study's participation.

SE21: Subject in a situation, which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

SE22: Subject not able to understand and/or to answer to the questions. SE23: Athletes as defined as routinely performing strenuous daily exercise for more than 1.5 hours at a time.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gastro-intestinal symptoms are mostly reported in women subjects than in men.
Enrollment: 486 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Comparison between groups of scores of Digestive Symptoms Frequency Questionnaire (DSFQ) during 28 days of investigational product consumption (the higher the score, the more severe are the symptoms, min:0, no symptom, max:16). | From Baseline to Visit 4 (28 days).

SECONDARY OUTCOMES:
Comparison between groups of scores of Digestive Symptoms Frequency Questionnaire (DSFQ) during 28 days of investigational product consumption (the higher the score, the more severe are the symptoms, min:0, no symptom, max:16). | From Baseline to each weekly evaluation visits (Week1 to Week 4) (4 weeks from baseline).
Comparison between groups of scores of Intestinal Gas Questionnaire (IGQ) during 28 days of investigational product consumption (the higher the score, the more severe are the symptoms, min:0). | From Week0 (V2) to each weekly evaluation visits (Week1 to Week4).
Comparison between groups of scores of Profile of Mood States questionnaire Short Form (POMS-SF) during 28 days of investigational product consumption (a scoring guide needs to be follow to interpreted). | From Week0 (V2) to Week2 (V3) and Week4 (V4).
Comparison between and within groups of total and living bacteria cells counts of B.lactis (method PMA-PCR) during 28 days of investigational product consumption and after 1 week following product consumption cessation. | Between Week0 (V2), Week2 (V3), Week4 (V4) and Week5 (V5).

OTHER OUTCOMES:
Comparison between and within groups of Food Frequency Questionnaire (FFQ) during 28 days of investigational product consumption (an algorithm will be used to assess quantity and quality of nutriment intake, developed by MS Nutrition company). | Between Week0 (V2) and Week4 (V4).
Comparison between groups of scores of Digestive Symptoms Frequency Questionnaire (DSFQ) during 28 days of investigational product consumption (the higher the score, the more severe are the symptoms, min:0, no symptom, max:16). | From Week0 (V2) to each weekly evaluation visits (Week1 to Week4).
  Scoring comparison (no unit)
Comparison between groups of scores of Intestinal Gas Questionnaire (IGQ) during 28 days of investigational product consumption (the higher the score, the more severe are the symptoms, min:0). | From Week0 (V2) to each weekly evaluation visits (Week1 to Week4).
  Scoring comparison (no unit)
Exploratory endpoint: Comparison within and between groups of microbiota alpha diversity (metagenomic and metatranscriptomic to be defined) during 28 days study product consumption and after 1 week following product consumption cessation. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within and between groups of microbiota beta diversity (metagenomic and metatranscriptomic to be defined) during 28 days of study product consumption and after 1 week following product consumption cessation. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within and between groups of microbiota taxonomy (metagenomic and metatranscriptomic to be defined) during 28 days of study product consumption and after 1 week following product consumption cessation. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within and between groups of microbiota beta activity (metagenomic, analysis methods to be defined) during 28 days of investigational product consumption and after 1 week following product consumption cessation. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within and between groups of microbiota beta activity (metatranscriptomic, analysis methods to be defined) during 28 days of investigational product consumption and after 1 week following product consumption cessation. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within B.lactis group of microbiota alpha and beta-diversity (bioinformatic) during and following cessation of product consumption. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within B.lactis group of microbiota abundance (composition) (bioinformatic) during and following cessation of product consumption. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within B.lactis group of microbiota abundance (function, no specific method of measurement has been defined yet) during and following cessation of product consumption. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).
Exploratory endpoint: Comparison within B.lactis group of total and living bacteria cells counts of B.lactis (method PMA-PCR) during and following cessation of product consumption. | From Week0 (V2) to Week2 (V3), Week4 (V4), and Week5 (V5).

CONTACTS AND LOCATIONS:
Overall Officials: Rim HASSOUNA, PhD, Study Chair — Danone Research, Palaiseau, France
Locations (1):
- CEN Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No